CLINICAL TRIAL: NCT01808079
Title: A Genome-Wide Association Study in Wilms Tumor
Brief Title: Gene Analysis in Studying Susceptibility to Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN09B1; NCI-2013-00120 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN09B1; AREN09B1 (Other: Childrens Oncology Group); AREN09B1 (Other: CTEP)
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Recurrent Childhood Kidney Neoplasm; Stage I Kidney Wilms Tumor; Stage II Kidney Wilms Tumor; Stage III Kidney Wilms Tumor; Stage IV Kidney Wilms Tumor
MeSH Terms: conditions — Wilms Tumor

GROUPS / COHORTS (1):
- Ancillary-correlative (genetic markers of Wilms tumor): Samples are analyzed for SNP profiling using real-time PCR and MLPA.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies gene analysis in studying susceptibility to Wilms tumor. Finding genetic markers for Wilms tumor may help identify patients who are at risk of relapse.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To use a genome-wide association analysis to identify novel genetic variants that confer susceptibility to Wilms tumor.

II. To improve our understanding of the genetic architecture and etiology of Wilms tumor.

III. To facilitate the identification of genetic markers that are associated with an increased risk of developing of Wilms tumor and/or those at risk of aggressive disease, relapse, additional tumors and/or cancer in their offspring.

OUTLINE:

Samples are analyzed for single nucleotide polymorphism (SNP) profiling using real-time polymerase chain reaction (PCR) and multiplex ligation-dependent probe amplification (MLPA).

ELIGIBILITY:
Inclusion Criteria:

* 3000 samples from the 1958 Birth Cohort (58C) and 3000 from the UK Blood Service control series (NBS)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tissue Bank
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Frequencies between cases and controls at each SNP | Baseline
  Compared using the Cochran Armitage trend test (1-df). The data will be analyzed individually for the UK/US study populations and combined using a Mantel-Haenszel analysis adjusting for study group, and related methods which allow for different effects in each population (for confirmed loci, we will compare effects across populations).
Frequency of maternal and paternal allelic transmission for risk alleles | Baseline
  Compared using a chi-squared test.
Genetic variation on sub-phenotypes such as age at diagnosis, unilateral or bilateral disease, sex, and ethnicity | Baseline
Interactions between genetic variation and treatment success or prognosis | Baseline
Interactions between germline genetic variation and tumor phenotypes | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul Grundy, Principal Investigator — Children's Oncology Group
Locations (1):
- Childrens Oncology Group, Philadelphia, Pennsylvania, United States